CLINICAL TRIAL: NCT04943744
Title: Monitoring Gastrointestinal Responses In Food Oral Immunotherapy Using the Esophageal STRING Test
Brief Title: Gastrointestinal STRING Test With Oral Immunotherapy
Acronym: STRING
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Parent study closed to enrollment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Medical Director, Clinical Research Uni, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 58997
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Eosinophilic Disorder; Food Allergy
MeSH Terms: conditions — Eosinophilia; Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: This STRING companion study will examine markers of esophageal inflammation during the COMBINE study using a minimally-invasive testing device, the esophageal string test (EST). If participants of COMBINE consent to this companion study, they will undergo an esophageal string test at the following time points in COMBINE:
  * During screening, prior to week 0, which will be baseline for the STRING esophageal test
  * Week 8, After the 8 weeks of treatment with omalizumab/placebo
  * If dose-related gastrointestinal (GI) side effects occur during the week 10-32 treatment period (OIT and dupilumab/placebo)
  * At Week 32, after 24 weeks of treatment with OIT and dupilumab or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- String Test-cohort A (Other): Participants in the COMBINE study will have an EST performed at pre- specified timepoints (screening, week 8, and week 32) and as needed depending on GI symptoms.
  A. Omalizumab for 8 weeks followed by mOIT with placebo for dupilumab for 24 weeks (Cohort A: Omalizumab-facilitated mOIT)
  Interventions: Device: Entero-tracker; Biological: omalizumab
- String Test-cohort B (Other): Participants in the COMBINE study will have an EST performed at pre- specified timepoints (screening, week 8, and week 32) and as needed depending on GI symptoms.
  B. Omalizumab for 8 weeks followed by mOIT with dupilumab for 24 weeks (Cohort B: Omalizumab-facilitated mOIT with concurrent dupilumab)
  Interventions: Device: Entero-tracker; Biological: omalizumab; Biological: dupliumab
- String Test-cohort C (Other): Participants in the COMBINE study will have an EST performed at pre- specified timepoints (screening, week 8, and week 32) and as needed depending on GI symptoms.
  C. Placebo for omalizumab for 8 weeks followed by mOIT with dupilumab for 24 weeks (Cohort C: mOIT with concurrent dupilumab)
  Interventions: Device: Entero-tracker; Biological: dupliumab

INTERVENTIONS:
Device: Entero-tracker — Esophageal STRING test (Entero-tracker)
Biological: omalizumab — Used in the parent study
  Arms: String Test-cohort A; String Test-cohort B
Biological: dupliumab — Used in the parent study
  Arms: String Test-cohort B; String Test-cohort C

SUMMARY:
This STRING study will examine markers of esophageal inflammation using a minimally-invasive testing device, the esophageal string test (EST). The primary objective is to determine the effect of omalizumab (Xolair) and dupilumab (Dupixent) on markers of eosinophilic inflammation in the esophagus of subjects treated with omalizumab-facilitated mOIT(mult-allergen oral immunotherapy) and/or mOIT with concurrent dupilumab.

DETAILED DESCRIPTION:
This is a companion study to a phase 2 randomized, controlled, double-blind clinical trial using biologics to improve multi-allergen oral immunotherapy (mOIT) outcomes. The parent study (COMBINE NCT03679676) consists of a screening period, 8 weeks of omalizumab or placebo injections, and 24 weeks of OIT with dupilumab or placebo injections followed by an off-treatment period.

This STRING companion study will examine markers of esophageal inflammation during the COMBINE study using a minimally-invasive testing device, the esophageal string test (EST). If participants of COMBINE consent to this companion study, they will undergo an esophageal string test at the following time points in COMBINE:

* During screening, prior to week 0, which will be baseline for the STRING esophageal test
* Week 8, After the 8 weeks of treatment with omalizumab/placebo
* If dose-related gastrointestinal (GI) side effects occur during the week 10-32 treatment period (OIT and dupilumab/placebo)
* At Week 32, after 24 weeks of treatment with OIT and dupilumab or placebo

ELIGIBILITY:
Inclusion Criteria: • Participants, aged 5-55 years enrolled in the parent COMBINE trial

* Able to swallow the EST.

Exclusion Criteria: • Allergy to, or inability to ingest, gelatin

-

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of subjects with esophageal eosinophilia (EE) | 32 weeks
  (defined as an EST score ≥ 2.9) in subjects receiving omalizumab-facilitated mOIT and/or mOIT with concurrent

SECONDARY OUTCOMES:
Comparison of EST scores | 8 weeks
  Comparison of EST scores (composite measure of eosinophilic inflammation) before and after treatment with omalizumab

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chinthrajah, MD, Principal Investigator — Stanford University
Locations (1):
- Sean N Parker Center for Allergy and Asthma Research at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No